CLINICAL TRIAL: NCT05199363
Title: Pediatric Patient Experience on a Diagnostic Path
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Memorial Health Institute, Poland (Other)
Collaborators: Siemens Healthcare Sp. z o.o. (Unknown)
Responsible Party: Principal Investigator, Elżbieta Jurkiewicz, professor, Children's Memorial Health Institute, Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Nr510/2021_ChildrensMHIPoland
Record Dates: First submitted 2021-12-28; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Headache; Urinary Incontinence; Growth Deficiency; Visual Impairment; Psychomotor Retardation, Mild to Severe; Demyelinating Diseases; Brain Tumor
Keywords: child; magnetic resonance imaging; anxiety; patient experience
MeSH Terms: conditions — Headache; Urinary Incontinence; Vision Disorders; Psychomotor Disorders; Demyelinating Diseases; Brain Neoplasms; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Study participants will be randomly assigned into one of 4 groups:
  * Group A, 25% of the sample - patients subject to intervention No 1: "Information leaflet"
  * Group B, 25% of the sample - patients subject to intervention No. 2: "Educational movie"
  * Group C, 25% of the sample - patients subject to intervention No. 3 "Demonstration"
  * Group D, 25% of the sample - control group, with no intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Information leaflet (Active Comparator): Before examination study participant will obtain an information leaflet which includes descriptive and illustrative sections "Information for young patients and their caregivers. What is Magnetic Resonance Imaging and what is the examination like?"
  Interventions: Other: Information leaflet
- Educational movie (Active Comparator): Before examination study participant will be shown educational video with an radiology technologist and actors who role play the examination "What is MRI and what is the examination like?"
  Interventions: Other: Educational movie
- Demonstration (Active Comparator): Before examination study participant will take a part in scenario-based demonstration with the use of props such as the scanner model and a multimedia presentation "Scenario for a demonstration before a Magnetic Resonance examination for young patients and their caregivers".
  Interventions: Other: Demonstration
- Control (No Intervention): Study participant will obtain standard information about magnetic resonance imaging before examination.

INTERVENTIONS:
Other: Information leaflet — Before examination study participant will obtain an information leaflet which includes descriptive and illustrative sections "Information for young patients and their caregivers. What is Magnetic Resonance Imaging and what is the examination like?"
  Arms: Information leaflet
Other: Educational movie — Before examination study participant will be shown educational video with an radiology technologist and actors who role play the examination "What is MRI and what is the examination like?"
  Arms: Educational movie
Other: Demonstration — Before examination study participant will take a part in scenario-based demonstration with the use of props such as the scanner model and a multimedia presentation "Scenario for a demonstration before a Magnetic Resonance examination for young patients and their caregivers"
  Arms: Demonstration

SUMMARY:
The trial will determine the impact of an information- and education-focused interventions on the anxiety levels, and patients' experiences as well as satisfaction of patients aged 10-14 and their caregivers during the MR examination.

DETAILED DESCRIPTION:
The aims of the trial

1. Examining the level of anxiety of individuals undergoing magnetic resonance imaging (MRI) as patients or caregivers (anxiety is measured at two points: before and after the MRI procedure).

2. Examining subjective patients' and caregivers' assessments of the key factors which make up the Patient Experience, i.e. the sum of all interactions which influence perceptions of the patients and their caregivers. The Patient Experience in this sense includes what is perceived, understood and remembered by the patient and their relatives in terms of:

* access to services and resources
* coordination and safety
* effectiveness of the services
* communication and education
* patient empowerment
* respect and dignity
* ensuring physical wellbeing
* ensuring psychological wellbeing
* environment and comfort and consequent levels of satisfaction. The full set of factors will only be examined for the patients' caregivers, while for the patients themselves the set of factors will be limited to those which can be competently assessed by persons aged 10-14 years.

  3. Examining the extent to which education- and information-focused interventions, using a variety of media (information leaflets, educational video, demonstration with props), impact anxiety levels, individual elements of the experience, and patients' and caregivers' satisfaction levels.

  4. Examining the extent to which educational- and informational-focused interventions can increase patients' co-operation and thus contribute to shorter examination times (avoidance of repetition of sequences) and a reduction in the rate of interrupted examinations.
  1. The participants will be recruited by the registration staff of the Magnetic Resonance (MR) Laboratory from those enrolled for magnetic resonance examinations for clinical indications. It will be done during a routine reminder of the upcoming examination date. The staff member informs the patient's caregiver of a possibility to participate in the examination and, after obtaining a preliminary declaration of participation, of the necessity to arrive 1 hour before the predetermined time.
  2. When the patient and their caregiver arrive at the Registration of the Magnetic Resonance Laboratory, a registration staff member hands over the "Information on the Trial regarding the Paediatric Patient Experience on the Diagnostic Pathway" which contains details of the objectives, design, scope and duration of the procedures and inconvenience of the trial which will be conducted, the expected benefits to participants of the trial which is a research experiment, and the health risks and hazards for the participants, the arrangements regarding handling any adverse events, the measures undertaken to ensure respect for the participants' privacy and the confidentiality of their personal data, and the rules for access to relevant information concerning the participants obtained during implementation of the experiment and the overall results thereof and for further use of the results thereof. The investigator also informs the participants of the possibility of withdrawing from the trial at any stage, of the rules on compensation in the event of any harm and of the source of funding of the medical experiment. After answering any questions from the subject, the investigator collects a signed Informed Consent Form from both the caregiver and the child, together with the information about the trial attached to it.
  3. A staff member of the Registration of the Magnetic Resonance Laboratory draws an allocation to one of the Groups (A/B/C/D) from a pool of sealed envelopes together with a unique code for the trial and enters the code into all questionnaires used in the trial.
  4. An radiology technologist or psychologist (after receiving training in the objectives, protocol and tools of the trial) provides the interventions as they are appropriate to groups:

     * to Group A: the investigator gives the information leaflet "Information for young patients and their caregivers. What is MRI and what is the examination like?" and ensures that the patient and caregiver read it.
     * to Group B: the investigator plays the educational video "What is an MRI and what is the examination like?" to the patient and caregiver and ensures that the patient and caregiver familiarise themselves with it.
     * to Group C: the investigator conducts a scenario-based demonstration using props in the form of a model scanner and a multimedia presentation ("Scenario for demonstration before a magnetic resonance examination for young patients and their caregivers")." No intervention is carried out in Group D.
  5. The patient's caregiver completes the State-Trait Anxiety Inventory (STAI) questionnaire.
  6. The patient (assisted by a technician or psychologist) completes the State-Trait Anxiety Inventory for Children (STAIC) form.
  7. A standard process of preparing for the magnetic resonance examination by a technician follows, and the magnetic resonance examination is performed as clinically indicated.
  8. The technician completes the questionnaire entitled "Assessment of the patient's and their caregiver's cooperation during magnetic resonance examination".
  9. The caregiver again completes the State-Trait Anxiety Inventory (STAI) questionnaire.
  10. The patient's caregiver completes the questionnaire "Assessment of the experience of the patient's caregiver during magnetic resonance examination".
  11. The patient (assisted by a technician or psychologist) again fills in the "State-Trait Anxiety Inventory for Children (STAIC) questionnaire.
  12. The patient (assisted by a technician or psychologist) fills in the questionnaire "Evaluation of the patient's experience during the magnetic resonance examination".

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 10-14 years.
* Referred for magnetic resonance imaging due to clinical indications.
* Patients undergoing magnetic resonance examination for the first time.
* Possibility of cooperating with the patient during the examination, no need for sedation.
* Consent of the patients' caregivers to participate in the examination; in the case of patients ≥ 13 years of age, also the patients' consents.
* Absence of contraindications to magnetic resonance imaging

Exclusion Criteria:

* Lack of parental or patient consent to participate in the trial.
* Contraindications to undergo magnetic resonance imaging.
* Lack of possibility to cooperate with the patient during the examination and/or the need for general anaesthesia for the MR examination.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory for Children | through study completion, an average of 1 year
  Change in State-Trait Anxiety Inventory for Children score; minimum score=20, maximum score=60, higher scores mean a worse outcome

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory | through study completion, an average of 1 year
  Change in parent's State-Trait Anxiety Inventory score; minimum score=20, maximum score=80, higher scores mean a worse outcome

OTHER OUTCOMES:
Patient's experience questionaire | through study completion, an average of 1 year
  Questionaire which assesses patient's experience during Magnetic Resonance examination; minimum score=0, maximum score=10, higher scores mean a better outcome
Patient's caregiver/parent experience questionaire | through study completion, an average of 1 year
  Questionaire which assesses patient's caregiver experience during MR examination; minimum score=0, maximum score=10, higher scores mean a better outcome
Patient's and caregiver's co-operation during the MR examination questionaire | through study completion, an average of 1 year
  Questionnaire which assesses the level of co-operation with the patient and their caregiver; minimum score=0, maximum score=10, higher scores mean a better outcome; as well as the occurrence of certain phenomena such as the need for additional sequences or the need to interrupt the examination: no / yes, yes is a worse outcome (to be completed by the technician)

CONTACTS AND LOCATIONS:
Overall Officials: Elżbieta Jurkiewicz, MD, PhD, Principal Investigator — CMHI
Locations (1):
- Children Memorial Health Institute (CMHI), Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Makanjee CR, Bergh AM, Hoffmann WA. Healthcare provider and patient perspectives on diagnostic imaging investigations. Afr J Prim Health Care Fam Med. 2015 May 20;7(1):801. doi: 10.4102/phcfm.v7i1.801. PMID 26245604
- [Background] Carlsson S, Carlsson E. 'The situation and the uncertainty about the coming result scared me but interaction with the radiographers helped me through': a qualitative study on patients' experiences of magnetic resonance imaging examinations. J Clin Nurs. 2013 Nov;22(21-22):3225-34. doi: 10.1111/jocn.12416. PMID 24118524
- [Background] Munn Z, Pearson A, Jordan Z, Murphy F, Pilkington D, Anderson A. Addressing the Patient Experience in a Magnetic Resonance Imaging Department: Final Results from an Action Research Study. J Med Imaging Radiat Sci. 2016 Dec;47(4):329-336. doi: 10.1016/j.jmir.2016.04.007. Epub 2016 Jun 27. PMID 31047258
- [Background] Bolderston A. Patient Experience in Medical Imaging and Radiation Therapy. J Med Imaging Radiat Sci. 2016 Dec;47(4):356-361. doi: 10.1016/j.jmir.2016.09.002. Epub 2016 Oct 15. PMID 31047261
- [Background] Jensen JD, Allen L, Blasko R, Nagy P. Using Quality Improvement Methods to Improve Patient Experience. J Am Coll Radiol. 2016 Dec;13(12 Pt B):1550-1554. doi: 10.1016/j.jacr.2016.09.005. PMID 27888940